CLINICAL TRIAL: NCT06945289
Title: Efficacy of Let's Know! for Improving Oral Language in First Grade Students
Brief Title: Efficacy of Let's Know! First Grade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, R.J. Risueño, Principal Investigator, Arizona State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020398
Record Dates: First submitted 2024-12-12; First posted 2025-04-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Developmental Language Disorder and Language Impairment
Keywords: developmental language disorder; language intervention
MeSH Terms: conditions — Language Development Disorders; Language Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 2 units of a multicomponent intervention to improve vocabulary, text structure knowledge, inferencing, and comprehension monitoring within narrative and expository texts.
  Interventions: Behavioral: Let's Know!

INTERVENTIONS:
Behavioral: Let's Know! — This intervention is modified from a whole-classroom intervention by LARRC, 2018 and modified by Hogan et al. used in a larger NIH R01 investigation. We are examining the efficacy of the first two units used by Hogan et al.

SUMMARY:
Oral language skills are vital for reading comprehension. Some children, however, are at increased risk for reading comprehension difficulties due to underlying oral language deficits. School-based interventions that target children's abilities to understand and produce spoken language have shown positive effects for improving language and reading comprehension of children with typical development and those at-risk for language disorders, so it is likely that they will benefit children with low oral language skills.

The purpose of this study is to examine the efficacy of a small-group intervention for improve language skills in first grade students with low oral language skills.

DETAILED DESCRIPTION:
Oral language skills, which consist of both lower-level (vocabulary and grammar) and higher-level skills (inferencing, comprehension monitoring, and text structure knowledge) are crucial for reading comprehension. Children with low oral language skills are at increased risk for negative academic outcomes due to their deficits in understanding and producing language. Multi-component interventions have shown positive effects for improving language comprehension and reading comprehension outcomes of children with typical development and at-risk for language and literacy disorders, and thus may benefit children with low oral language skills.

The purpose of this study is to examine the efficacy of Let's Know!, a small group multi-component intervention, for improving language comprehension skills in first-grade students with low oral language skills. A randomized controlled trial will be employed to compare the language comprehension outcomes for a treatment group compared to a business-as-usual control group.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in first-grade;
* receive a score of below than 5 on two items on the Student Language Scale (Nelson et al., 2018) or be receiving school speech-language services for language impairment;
* be proficient in English, per caregiver report;
* have no other neurological impairments (e.g., intellectual disability, autism) per parent report;
* have corrected vision;
* no hearing impairment.

Exclusion Criteria:

* cannot be enrolled in English-Language Learner services in the school.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Curriculum-Aligned Vocabulary Measure | From enrollment to the end of treatment at 10 weeks of intervention.
  Vocabulary measure to assess participants' knowledge of 16 vocabulary words taught during the intervention.
Curriculum-Aligned Inferencing Measure | From enrollment to the end of treatment at 10 weeks of intervention.
  This measure will examine students' knowledge of making inferences through narrative texts. There are 16 total questions for this measure.
Curriculum-Aligned Comprehension Monitoring Measure | From enrollment to the end of treatment at 10 weeks of intervention.
  This is a curriculum-aligned measure of comprehension monitoring strategies taught during intervention. There are 4 total questions for this measure.
Curriculum-Aligned Text Structure Knowledge Measure | From enrollment to the end of treatment at 10 weeks of intervention.
  This is a curriculum-aligned measure of text structure knowledge taught during the intervention. The participant is read a story, is asked to retell the story, and then is asked 3 questions about main events. This occurs twice for a total of 2 retells and 6 comprehension questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
In our parent consent form, we did not specify that individual participant data would be shared.